CLINICAL TRIAL: NCT06942286
Title: HPV DNA Screening With Self-Collection Method and Its Management in the Context of Population-Based Cervical Cancer Screening Pilot Project in Indonesia
Brief Title: Primary HPV Self-Collection in Indonesia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dharmais National Cancer Center Hospital (Other Government)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DP.04.03/11.10/041/2025
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancers; CIN - Cervical Intraepithelial Neoplasia; Human Papillomavirus (HPV)
Keywords: Human Papilomavirus (HPV); Cervical Cancer; Cervical Dysplasia; HPV Self-Collection; HPV Self-Sampling; Primary HPV Test
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HPV Self-Collection (Experimental): Participants will perform HPV self-collection.
  Interventions: Diagnostic Test: HPV Self-Collection

INTERVENTIONS:
Diagnostic Test: HPV Self-Collection — Participants will perform HPV self-collection.

SUMMARY:
The purpose of this study is to implement human papillomavirus (HPV) self-collection in Indonesia.

DETAILED DESCRIPTION:
After participants give informed consent, they will receive a short educational session about cervical cancer and HPV, after which they will be offered the opportunity to undergo primary HR-HPV testing via self-collection. Participants will be contacted within 4 weeks with their results. Those who test positive for high-risk HPV will receive a follow-up appointment, at which time visual assessment with acetic acid and/or colposcopy will be performed. Those with detectable lesions and/or HPV 16/18+ will undergo treatment with thermal ablation. If they are ineligible for thermal ablation, they will undergo cervical biopsy, endocervical curettage, and/or loop electrosurgical excision procedure (LEEP) as indicated. Anyone with suspicion for cancer will undergo biopsies and referral to a gynecologic oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-69 years old
* Have not had a Pap test within the last 3 years or an HPV test within the last 5 years
* Have never been diagnosed with cervical cancer or high-grade dysplasia
* Have no history of hysterectomy with cervical removal
* Expressed willingness to participate in the study, including conducting HPV self-collection, follow-up treatment, and related surveys

Exclusion Criteria:

* Being pregnant or within 6 weeks postpartum
* Women who have never engaged in sexual activity
* Medical, psychiatric, or other conditions that may interfere with compliance with protocols, security assessments, and/or ability/competence to give informed consent
* Adults who do not have the capacity to give consent may be excluded, as participants must be able to perform activities required by the protocol

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Success Rate of HPV Self-Collection | from enrollment to receipt of results, up to 8 weeks
  number of subjects with valid HPV test results from self-collection / number of eligible subjects

SECONDARY OUTCOMES:
HPV Self-Collection Invitation Coverage | from enrollment to receipt of results, up to 8 weeks
  number of subjects with valid HPV test results from self-collection / total eligible population in the catchment area
HPV Self-Collection Participation Rate | from enrollment to receipt of results, up to 8 weeks
  number of subjects with samples received at the laboratory / number of invited subjects
Examination Coverage of HPV Self-Collection | from enrollment to receipt of results, up to 8 weeks
  number of subjects with samples received at the laboratory / total eligible population in the catchment area
HPV Self-Collection Acceptance Rate | from enrollment to specimen collection, up to 2 weeks
  number of subjects who perform self-collection / number of subjects given HPV self-collection kits and instructions
Preference for HPV Self-Collection | from enrollment to specimen collection, up to 2 weeks
  number of subjects who choose self-collection / number of subjects who answered survey questions
Patient Follow-up Rate | from receipt of results to follow-up exam, up to 60 days
  number of subjects who receive VIA follow-up within 60 days / number of subjects with positive HPV tests

OTHER OUTCOMES:
HPV Test Validity | from specimen collection to receipt of results, up to 6 weeks
  number of valid HPV test results / number of HPV tests
Time from HPV Self-Collection to Receipt of Sample in Lab | from specimen collection to receipt of sample in laboratory, up to 2 weeks
  number of days from HPV self-collection until sample is received in the laboratory
Time from Receipt of Sample in Lab to Result Reporting | receipt of sample in laboratory to receipt of results, up to 4 weeks
  number of days from receipt of HPV sample in laboratory to availability of results
Time from Result Reporting to Patient Follow-up | from receipt of results to follow-up exam, up to 6 months
  number of days from result reporting to patient presenting for follow-up examination
Average Cycle Threshold Values by Genotype | from specimen collection to receipt of results, up to 6 weeks
  average cycle threshold value for each genotype in all subjects with a reportable cycle threshold value for that genotype

CONTACTS AND LOCATIONS:
Overall Officials: Widyorini L Hanafi, MD, Principal Investigator — Dharmais National Cancer Center Hospital; Dian T Sinulingga, MD, M.Epid, Principal Investigator — Dharmais National Cancer Center Hospital
Locations (3):
- Indonesia (3):
  - Puskesmas Lebak, Lebak, Banten
  - Dharmais National Cancer Center Hospital, Jakarta, Jakarta Special Capital Region
  - Puskesmas Depok, Depok, West Java

IPD SHARING:
Plan to Share IPD: No